CLINICAL TRIAL: NCT00695370
Title: Hematopoietic Progenitor Cell Mobilization in Children With Malignancies: Evaluation of Pegfilgrastim at 300µg/kg in Hematological Steady State
Brief Title: Evaluation of Pegfilgrastim for Stem Cell Mobilization in Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruiting or enrolling participants has halted and will not resume
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Amgen (Industry)
Responsible Party: Dr Etienne MERLIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0035
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Solid Malignancies
Keywords: Children; cancer; Bone marrow transplantation; Mobilization; G-CSF; Children with solid malignancies
MeSH Terms: conditions — Neoplasms | interventions — pegfilgrastim; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Pegfilgrastim (drug)

SUMMARY:
Hypothesis: pegfilgrastim at 300 µg/kg in hematological steady state provides an efficient stem cell mobilization in children with malignancies

Design: phase 2 study.

Judgment criterion: percentage of children achieving at least 5x10e6 CD34 cells with a standard apheresis (less than 2 blood volume processed)

DETAILED DESCRIPTION:
Patients: consecutively referred for HSC mobilization. At least 17 days after the previous chemotherapy. No hematological growth factor during the 8 previous days.

Mobilization: one sc injection of 300 µg/kg pegfilgrastim (Neulasta, Amgen)

Evaluation during the study: CD34 circulating cells from day 2 to day 7 ; AE recording

Judgment criterion: percentage of children achieving at least 5x10e6 CD34 cells with a standard apheresis (less than 2 blood volume processed)

Analysis: sequential Bayesian study

ELIGIBILITY:
Inclusion Criteria:

* 0 to 18 years
* solid malignancy
* Lansky score >70%
* more than 17 days since the beginning of the last chemotherapy cycle
* absolute neutrophil count (ANC) greater than 1×109/l
* no administration of any hematopoietic growth factor in the previous 8 days

Exclusion Criteria:

* clinical or biological conditions precluding the mobilization or collection procedure

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-12 (Estimated); Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
percentage of children achieving at least 5x10e6 CD34 cells with a standard apheresis (less than 2 blood volume processed)

SECONDARY OUTCOMES:
Side effects Number of apheresis required to achieved a graft of at least 5x10e6 CD34 cells

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Merlin, MD, Principal Investigator — University Hospital, Clermont-Ferrand